CLINICAL TRIAL: NCT02454400
Title: Pre-surgery Physiotherapy for Patients With Specific Low Back Pain , RCT
Brief Title: Pre-surgery Physiotherapy for Patients With Specific Low Back Pain
Acronym: PREPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Ostergotland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Birgitta Oberg, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prepare
Record Dates: First submitted 2015-04-29; First posted 2015-05-27 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Lumbar Spine Disc Herniation; Spinal Stenosis; Spondylolisthesis, Grade 4
Keywords: physical therapy; lumbar spine surgery; pre-surgical intervention; RCT
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-surgery physiotherapy (Other): Twice a week, in 9 weeks
  Interventions: Other: Pre-surgery physiotherapy
- Waiting-list (Other): Standard information by the orthopedic surgeon
  Interventions: Other: Waiting-list

INTERVENTIONS:
Other: Pre-surgery physiotherapy — Physiotherapy guided intervention twice a week for nine weeks. The program includes:
  1. Active physiotherapy according to a treatment based classification:
     1. Specific exercises and mobilization
     2. Motor control exercises
     3. Traction
  2. Tailor-made general supervised exercise program
  3. Behavioral approach to reduce fear avoidance and increase activity level.
  4. Standardized information about:
     1. the surgery
     2. post-surgery rehabilitation
     3. to stay active
  Arms: Pre-surgery physiotherapy
Other: Waiting-list — Standardized information about:
  1. the surgery
  2. post-surgery rehabilitation
  3. to stay active
  Arms: Waiting-list

SUMMARY:
The aim is to study if pre-surgery physiotherapy improves function, pain and health in patients with specific low back pain scheduled for surgery. Patients are followed over a two year period. A secondary aim is to study what factors predict short and long term outcomes.

DETAILED DESCRIPTION:
The design is a randomized controlled trial, where patients are allocated either to pre-surgery physiotherapy or waiting-list when scheduled for surgery due to specific low back pain (spinal stenosis, disc herniation, spondylolisthesis, disc degenerative disease (DDD)).

The patients are scheduled for surgery due to specific low back pain diagnosis and randomized to either pre-surgery physiotherapy or waiting-list group. Clinical measurement and treatment-classification is done before and after intervention.

Pre-surgery intervention:

Physiotherapy guided intervention twice a week for nine weeks. The program includes:

1. Active physiotherapy according to a treatment based classification

   1. Specific exercises and mobilization
   2. Motor control exercises
   3. Traction
2. Tailor-made general supervised exercise program
3. Behavioral approach to reduce fear avoidance and increase activity level.

Both groups receive standardized information about surgery, post-surgery rehabilitation and to stay active.

Surgery in performed according to existing guidelines.

Measurements:

Patients fill out a questionnaire at baseline, before surgery (after pre-surgery physiotherapy or waiting-list), three months, one and two years after surgery. The questionnaire includes self-reported measures for function Oswestry Disability Index (ODI) (primary outcome), pain (VAS, pain drawing, pain duration) and health (SF-36, EQ-5D), anxiety, depression (HADS), self efficacy, fear avoidance belief questionnaire (FABQ), workability, (WAI), expectations, general information of work, sick-leave, lifestyle behavior, previous healthcare consumption, patient reported treatment effects, patient enablement instrument (PEI), and adverse events.

Clinical measurement is done before and after intervention. Clinical measurements includes; isometric quadriceps strength, walking-test, neurological tests for L4-S1, SI-joint tests, Posterior-anterior-test (PA-test), test for centralization, test for aberrant movements.

ELIGIBILITY:
Inclusion Criteria:

Patients that are scheduled for surgery due to following diagnoses;

* Disc herniation,
* Spinal stenosis,
* Spondylolisthesis,
* Degenerative disc disease.
* Fluent in Swedish.

Exclusion Criteria:

* need of acute surgery
* other severe diagnoses.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2012-09; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Change in ODI from baseline to after intervention (after 3 months) and 3 months, 1 and 2 years post-surgery

SECONDARY OUTCOMES:
Visual analog scale for lumbar pain | Change in ODI from baseline to after intervention (after 3 months) and 3 months, 1 and 2 years post-surgery
  Self reported pain in lumbar and leg pain respectively
Visual analog scale for leg pain | Change in ODI from baseline to after intervention (after 3 months) and 3 months, 1 and 2 years post-surgery
  Self reported pain in lumbar and leg pain respectively
Health (SF-36, EQ-5D) | Change in ODI from baseline to after intervention (after 3 months) and 3 months, 1 and 2 years post-surgery
  Self reported health
Anxiety, depression (HADS) | Change in ODI from baseline to after intervention (after 3 months) and 3 months, 1 and 2 years post-surgery
  Self reported anxiety and depression
Self efficacy (SES) | Change in ODI from baseline to after intervention (after 3 months) and 3 months, 1 and 2 years post-surgery
  Self reported self efficacy
Fear avoidance belief questionnaire (FABQ) | Change in ODI from baseline to after intervention (after 3 months) and 3 months, 1 and 2 years post-surgery
  Self reported fear avoidance belief questionnaire
Workability, (WAI) | Change in ODI from baseline to after intervention (after 3 months) and 3 months, 1 and 2 years post-surgery
  Self reported workability

CONTACTS AND LOCATIONS:
Overall Officials: Birgitta Öberg, professor, Principal Investigator — Div Physiotherapy, department of Health and Science, Linkoping University
Locations (1):
- University Hospital, Linköping, Östergötland County, Sweden

REFERENCES:
- [Derived] Fors M, Enthoven P, Abbott A, Oberg B. Effects of pre-surgery physiotherapy on walking ability and lower extremity strength in patients with degenerative lumbar spine disorder: Secondary outcomes of the PREPARE randomised controlled trial. BMC Musculoskelet Disord. 2019 Oct 24;20(1):468. doi: 10.1186/s12891-019-2850-3. PMID 31651299
- [Derived] Lindback Y, Tropp H, Enthoven P, Abbott A, Oberg B. PREPARE: presurgery physiotherapy for patients with degenerative lumbar spine disorder: a randomized controlled trial. Spine J. 2018 Aug;18(8):1347-1355. doi: 10.1016/j.spinee.2017.12.009. Epub 2017 Dec 15. PMID 29253630
- [Derived] Lindback Y, Tropp H, Enthoven P, Abbott A, Oberg B. PREPARE: Pre-surgery physiotherapy for patients with degenerative lumbar spine disorder: a randomized controlled trial protocol. BMC Musculoskelet Disord. 2016 Jul 11;17:270. doi: 10.1186/s12891-016-1126-4. PMID 27400960